CLINICAL TRIAL: NCT05334927
Title: China HeadAche DIsorders RegiStry
Acronym: CHAIRS
Status: Recruiting | Type: Observational
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Yonggang.wang, MD, Beijing Tiantan Hospital
Other Study IDs: KY2022-tt02
Record Dates: First submitted 2022-01-20; First posted 2022-04-19 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2025-12

CONDITIONS: Headache Disorders, Primary; Migraine; New Daily Persistent Headache; Medication Overuse Headache; Tension-Type Headache; Trigeminal Autonomic Cephalalgia
MeSH Terms: conditions — Headache Disorders, Primary; Migraine Disorders; Headache Disorders, Secondary; Tension-Type Headache; Trigeminal Autonomic Cephalalgias | interventions — erenumab; eptinezumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Biospecimen Retention: Samples With DNA — Whole Blood;serum; Saliva; Feces; Urine; Cerebral Spinal Fluid
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Medicine Overuse Headache/New Daily Persistent Headache: The first 18 months were followed up once a month,then followed up once at the 24th month,follow-up visits were made annually after 24 months
  Interventions: Behavioral: Medicine Overuse Headache/New Daily Persistent Headache
- Chronic Migraine: The patients were followed up at 1, 2, 3, 6, 9, 12, 18 and 24 months,then follow-up visits were made annually
  Interventions: Behavioral: Episodic Migraine and Chronic Migraine; Drug: Yangxue Qingnao Granules (Pills); Biological: Erenumab; Biological: Eptinezumab
- Patients with other types of primary headache: The patients were followed up at 3, 6, 9months
  Interventions: Behavioral: Patients with other types of primary headache
- Episodic migraine: The patients were followed up at 1, 2, 3, 6, 9, 12, 18 and 24 months,then follow-up visits were made annually.
  Interventions: Drug: Yangxue Qingnao Granules (Pills); Biological: Erenumab; Biological: Eptinezumab

INTERVENTIONS:
Behavioral: Medicine Overuse Headache/New Daily Persistent Headache — At the end of the 24th month visit, the patient is free to choose whether to conduct a face-to-face visit once a year until death.
  Groups: Medicine Overuse Headache/New Daily Persistent Headache
Behavioral: Episodic Migraine and Chronic Migraine — long-term follow-up
  Groups: Chronic Migraine
Behavioral: Patients with other types of primary headache — No collection Brain imaging、Cognitive function test、Biological sample
  Groups: Patients with other types of primary headache
Drug: Yangxue Qingnao Granules (Pills) — Participants who, in routine clinical practice, were prescribed Yangxue Qingnao Granules/Pills for acute headache relief and/or preventive management were enrolled. Treatment initiation, dosing, frequency, and duration were determined by the treating physician and the patient and were not assigned by the study protocol. During the 12-week observation period, participants were followed and outcomes were recorded, including relief of up to four headache episodes (for those using the medication for acute treatment) and longitudinal symptom measures at weeks 4, 8, and 12 (for those receiving preventive management).
  Groups: Chronic Migraine; Episodic migraine
Biological: Erenumab — Participants who received eptinezumab for migraine prophylaxis in routine clinical practice were included. Treatment decisions (including whether to initiate eptinezumab, the selected dose [e.g., 100 mg or 300 mg], infusion interval, and duration) were made by the treating physician in consultation with the patient, and were not assigned by the study protocol. Patients were followed prospectively/retrospectively according to routine clinic visits, with outcome assessments captured at approximately 4-week intervals during the 12-week observation window (and additional follow-up when available).
  Groups: Chronic Migraine; Episodic migraine
Biological: Eptinezumab — Participants who received eptinezumab for migraine prophylaxis in routine clinical practice were included. Treatment decisions (including whether to initiate eptinezumab, the selected dose [e.g., 100 mg or 300 mg], infusion interval, and duration) were made by the treating physician in consultation with the patient, and were not assigned by the study protocol. Patients were followed prospectively/retrospectively according to routine clinic visits, with outcome assessments captured at approximately 4-week intervals during the 12-week observation window (and additional follow-up when available).
  Groups: Chronic Migraine; Episodic migraine

SUMMARY:
It is planned to include 10000 patients. In the China HeadAche DIsorders RegiStry CHAIRS）, patients aged over 12 years with primary headache and medication-overuse headache(MOH) were collected. The biomarkers, imaging features, cognition, genetic characteristics, ocial and demographic data, medical data, therapeutics used, and outcome of headache-related diseases were studied, and long-term follow-up was planned.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 12 years old,Any gender;
2. The first onset age of primary headache was less than 50 years old(Age <65 years at first diagnosis of chronic migraine);
3. patients with primary headache (migraine, tension headache and other types of primary headache) or primary headache complicated with MOH according to ICHD-3;
4. Sign the informed consent form.

Exclusion Criteria:

1. According to the ICHD-3 diagnostic criteria, there are still headaches directly related to secondary factors (except drug overuse) at the time of enrollment;
2. Those who cannot be diagnosed as primary headache or primary headache combined with medication overuse headache according to ICHD-3;
3. According to DSM-V diagnostic criteria, patients with severe mental diseases (such as schizophrenia, mental disorders associated with mental retardation, etc.);
4. Patients with severe organic diseases, such as malignant tumors, and the expected survival time is less than 1 year;
5. Pregnant,planning pregnancy or Lactating women;
6. Subjects participating in other clinical trials;
7. Unable to cooperate to complete the follow-up due to geographical or other reasons

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with primary headache (migraine, tension headache and other types of primary headache) or primary headache complicated with MOH according to ICHD-3.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2022-08-29 (Actual); Primary Completion 2031-12-31 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
Headache Days | long term: 10 years
  The number of days of headache is the number of days in which headache occurs.
MRI change | long term: 10 years
  Patients will accept MRI scans will be done at baseline and once per year.
Genetic analysis of familial headache | 1 year
  Blood samples will be collected from all participants who consent to participate in the study, for the purposes of genetic analysis of familial headache.
Montreal Cognitive Assessment (MoCA) | long term: 10 years
  The Montreal Cognitive Assessment (MoCA) will be used to assess changes in cognitive functions.
Mini-Mental State Exam (MMSE) | long term: 10 years
  The Mini-Mental State Examination (MMSE) is a 30-point questionnaire that is used in clinical and research settings to assess cognitive function.
Migraine Disability Assessment (MIDAS) | long term: 10 years
  The MIDAS is a 7-item questionnaire designed to quantify headache-related disability over a 3- month period. The MIDAS score is the sum of missed work or school days, days at work or school plus days of household work where productivity was reduced by half or more, missed household work days, and missed non-work activity days due to headaches in the last 3 months.
Generalized Anxiety Disorder (GAD-7) | long term: 10 years
  GAD-7 is a proven, self-administered and concise tool for screening and diagnosing mental health disorders, which has been tested in the field in office practice. The GAD-7 scale score ranges from 0 to 21.
Patient Health Questionnaire (PHQ)-9 | long term: 10 years
  The PHQ-9 is the depression module, which scores each of the 9 DSM-IV criteria as "0" (not at all) to "3" (nearly every day). A PHQ-9 score total of 0-4 points equals "normal" or minimal depression. Scoring between 5-9 points indicates mild depression, 10-14 points indicates moderate depression, 15-19 points indicates moderately severe depression, and 20 or more points indicates severe depression.
Pain freedom at 2 hours | 2 hours post-dose
  It refers to the complete resolution of headache symptoms within 2 hours after taking the investigational drug, without the use of any rescue medication, and without recurrence of headache during this period.

SECONDARY OUTCOMES:
Social and demographic data, medical history | long term: 10 years
  Social and demographic data, medical and medication history will be collected at initial screening.
Use of Rescue Medication | long term: 10 years
  Frequency of Rescue medication will be collected by eDiary.
Moderate / Severe Headache Days | long term: 10 years
  Moderate / severe headache days are defined as a day in which moderate or severe pain persists for at least 4 hours, or headache lasts for one day after successful medication for acute headache. These definitions allow the use of relatively simple headache diaries. Subjects were required to indicate whether headache was present (yes / no), peak (mild / moderate / severe) severity and duration (< 4h or 4h), type of acute drug intake, and response to treatment should also be recorded.
Pain severity | long term: 10 years
  Pain severity were captured through Visual analogue scale (VAS) for pain, a continuous scale comprised of a horizontal line, anchored by "no pain" (score of 0) and "worst imaginable pain" (score of 10).
MEG | long term: 10 years
  Patients will accept MEG.
PET | long term: 10 years
  Patients will accept PET scan.
EEG | long term: 10 years
  Patients will accept EEG scan.
Proteomics | 1 year
  Blood, urine and Cerebrospinal fluid samples will be collected from all participants who consent to participate in the study, for the purposes of Proteomics at baseline and month 12.
Microbiome | 1 year
  Saliva samples will be collected from all participants who consent to participate in the study, for the purposes of Microbiome at baseline and month 12.
Headache Impact Test (HIT-6) | long term: 10 years
  The HIT-6 is a 6-question assessment used to measure the impact headaches have on a participant's ability to function on the job, at school, at home, and in social situations. It assesses the effect that headaches have on normal daily life and the participant's ability to function.
European Quality of Life 5 Dimensions 3 Level Version (EQ-5D-3L) | long term: 10 years
  EQ-5D-3L is a generic instrument for use as a measure of health status. The EQ-5D-3L consists of 2 components-the EQ-5D descriptive system and the EQ VAS. The descriptive system comprises of 5 dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression). The respondent is asked to indicate his/her health state by ticking (or placing a cross) in the box against the most appropriate statement in each of the 5 dimensions.
  The EQ VAS records the respondent's self-rated health on a vertical, VAS where the endpoints are labelled "Best imaginable health state" and "Worst imaginable health state." The scoring range of the EQ VAS is from 0 (worst imaginable health) to 100 (best imaginable health).
Migraine Specific Quality of Life Questionnaire, Version 2.1 (MSQ v2.1) | long term: 10 years
  The MSQ v2.1 is a 14-item questionnaire designed to measure health-related quality-of-life impairments attributed to migraine in the past 4 weeks. It is divided into 3 domains: Role Function Restrictive assesses how migraines limit one's daily social and work-related activities; Role Function Preventive assesses how migraines prevent these activities; and the Emotional Function domain assesses the emotions associated with migraines.
Pittsburgh Sleep Quality Index (PSQI) | long term: 10 years
  The Pittsburgh Sleep Quality Index (PSQI) is an effective instrument used to measure the quality and patterns of sleep.
Columbia-Suicide Severity Rating Scale | long term: 10 years
  C-SSRS will be administered to study subjects at each study visit to assess possible suicidal ideation and behavior. Reports of suicidal ideation with intent to act (endorse item 4 or 5) and reports of actual, aborted, or interrupted suicide attempts or a behavior preparatory for making an attempt indicate subjects at high risk for suicide.
Absence of the most bothersome symptom | 2 hours post-dose
  It refers to the complete resolution of the patient's self-identified most bothersome migraine-associated symptom (including photophobia, phonophobia, nausea, etc.) within 2 hours after taking the study medication.
Patient Global Impression of Change (PGIC) Scale | 10 years
  The Patient Global Impression of Change (PGIC) Scale is a single-item, patient-reported measure of overall change in symptoms, activity limitation, mood, and overall quality of life since starting treatment at this institution. Scores range from 1 to 7, where 1 = no improvement (or condition worsened) and 7 = very large improvement; higher scores indicate better improvement (better outcome).
Fatigue Impact Scale (FIS) | 10 years
  Fatigue Impact Scale (FIS) is a standardized questionnaire assessing the impact of fatigue on daily functioning (cognitive, physical, and psychosocial domains). Each item is scored 0-4; the total score ranges from 0 to 160 (sum of 40 items). Higher scores indicate greater fatigue impact (worse outcome).

CONTACTS AND LOCATIONS:
Locations (20):
- China (20):
  - Beijing Tiantan Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing Chaoyang Hospital, Beijing, Beijing Municipality
  - Chongqing People's Hospital, Chongqing, Chongqing Municipality
  - Fujian Provincial Hospital, Fuzhou, Fujian
  - The First Affiliated Hospital of Guangxi University of Chinese Medicine, Nanning, Guangxi
  - The First People's Hospital of Zunyi, Zunyi, Guizhou
  - Ruijin-Hainan Hospital Shanghai Jiao Tong University School Of Medicine, Qionghai, Hainan
  - Zhangjiakou First Hospital, Zhangjiakou, Hebei
  - Luohe Central Hospital, Luohe, Henan
  - Luoyang Central Hospital, Luoyang, Henan
  - The Second Affiliated Hospital of Henan University of Science and Technology, Luoyang, Henan
  - The 7th People's Hospital of Zhengzhou, Zhengzhou, Henan
  - Changzhou First People's Hospital, Changzhou, Jiangsu
  - Jiujiang First People's Hospital, Jiujiang, Jiangxi
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Huludao Central Hospital, Huludao, Liaoning
  - Zibo Municipal Hospital, Zibo, Shandong
  - Dachuan District People's Hospital, Dazhou, Sichuan
  - Deyang People's Hospital, Deyang, Sichuan
  - The First People's Hospital of Guangyuan, Guangyuan, Sichuan

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: CSR

REFERENCES:
- [Derived] Xiong Z, Qiu D, Liang J, Li X, Guo Z, Zhang M, Liu G, Gao T, Wang Y. Disrupted functional network topology in tension-type headache: A cross-sectional magnetoencephalography study. Cephalalgia. 2025 Oct;45(10):3331024251386425. doi: 10.1177/03331024251386425. Epub 2025 Oct 15. PMID 41091912
- [Derived] Wang W, Qiu D, Mei Y, Bai X, Yuan Z, Zhang X, Xiong Z, Tang H, Zhang P, Zhang Y, Yu X, Wang Z, Ge Z, Sui B, Wang Y. Altered functional connectivity of brainstem nuclei in new daily persistent headache: Evidence from resting-state functional magnetic resonance imaging. CNS Neurosci Ther. 2024 Mar;30(3):e14686. doi: 10.1111/cns.14686. PMID 38516817
- [Derived] Wang W, Yuan Z, Zhang X, Bai X, Tang H, Mei Y, Qiu D, Zhang Y, Zhang P, Zhang X, Zhang Y, Yu X, Sui B, Wang Y. Mapping the aberrant brain functional connectivity in new daily persistent headache: a resting-state functional magnetic resonance imaging study. J Headache Pain. 2023 Apr 26;24(1):46. doi: 10.1186/s10194-023-01577-2. PMID 37098469